CLINICAL TRIAL: NCT06141551
Title: Intradural Disc Herniation: a Case Report and Review of Complications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gansu Provincial Hospital (Other)
Responsible Party: Principal Investigator, ZhenHu, doctor-in-charge, Gansu Provincial Hospital
Other Study IDs: CR20231001
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Disc Herniation
Keywords: Intradural disc herniation; Complications; Degenerative spinal disease; Decompression
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: total laminectomy decompression — Surgical decompression
  Other Names: posterior approach lumbar spinal fusion

SUMMARY:
This observational study collects clinical data as well as pathological reports from a patient with an intradural disc herniation, reports on the course of the patient's recovery through surgical treatment, summarizes the complications of this type of disease, and provides new ideas for improving the chances of preoperative diagnosis.

DETAILED DESCRIPTION:
We collect the patient's personal history, family history, reason for visit, visit flow, clinical data, pathology reports, and surgical images and videos.

ELIGIBILITY:
Inclusion Criteria:

* IDH patients

Exclusion Criteria:

* no

Ages: 40 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: A male 40-year-old patient with IDH
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
physiology | 07/2023
  Grayish-white tissue identified as degenerated disc tissue was removed from the patient's lumbar spine partially within the dura mater

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, Dr, Study Director — Gansu Provincial People's Hospital
Locations (1):
- Gansu Provincial People's Hospital, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
The patients in this study rejected this